CLINICAL TRIAL: NCT06541847
Title: A Phase 2, Open-Label, Single Arm, Non-Controlled, Single-Stage Study to Evaluate the Safety and Effects of HLX-1502 in Patients With Plexiform Neurofibroma and Neurofibromatosis Type 1
Brief Title: A Phase 2, Open-Label Study to Evaluate the Safety and Effects of HLX-1502 in Patients With Neurofibromatosis Type 1
Acronym: INSPIRE-NF1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Healx Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX015-0201
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Neurofibromatosis Type 1
Keywords: Neurofibromatosis Type 1; Plexiform Neurofibroma; pediatric
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HLX-1502 (Experimental): Participants will take an oral dose three times a day (with or without food) for 12 cycles. A cycle is defined as 28 days. Participants with a partial response or stable disease with a previously progressive tumor and/or clinical improvement can continue therapy for an additional 12 cycles for a total of 24 cycles.
  Interventions: Drug: HLX-1502

INTERVENTIONS:
Drug: HLX-1502 — Participants will take an oral dose three times a day (with or without food) for up to 24 cycles (a cycle is defined as 28 days).

SUMMARY:
The trial will be an open label, single arm, phase 2 study to assess the tolerability and efficacy of HLX-1502 in participants with NF1 that are 16 years or older in age with progressive and/or symptomatic PN. This study will also investigate the safety and efficacy of HLX-1502 in a small cohort of 12 to 15 year olds.

ELIGIBILITY:
Inclusion Criteria:

1. All participants must have a diagnosis of NF1 based on the 2021 revised consensus criteria.
2. Participants must have PN(s) that are progressive OR are causing significant morbidity, such as (but not limited to) head and neck lesions that are compromising the airway or great vessels, brachial or lumbar plexus lesions that are causing nerve compression and loss of function, lesions causing significant disfigurement (e.g., orbital lesions), lesions of the extremity that cause limb hypertrophy or loss of function, and painful lesions. Participants with paraspinal PN will be eligible for this trial. Histologic confirmation of tumor is not necessary but should be considered if there are clinical or radiographic findings concerning for malignant transformation of a PN.
3. Measurable Disease: Participants must have measurable PN(s) amenable to volumetric MRI analysis. For the purpose of this study, the target lesion must be seen on at least 3 consecutive MRI slices and the field of view must contain the entire tumor of interest. Tumors must be at least 3 mL in volume (most PN 3 cm in longest diameter will meet this criteria). If the tumor is < 3 cm in longest diameter, the participant may still be eligible. Central review of the MRI of the target PN is required prior to enrollment to ensure that the tumor is measurable and amenable to volumetric analysis.
4. Age: Participants must be ≥ 12 years of age at the time of study entry. Note: Although prior MEKi therapy is not a requirement, patients should be counseled on the availability of FDA-approved MEKi therapies prior to enrollment.
5. Weight ≥ 42 kg.
6. Performance Level: Participants must have a Lansky (12-15 years of age) or Karnofsky (16+ years of age) score ≥ 50%.
7. Organ Function Requirements: Adequate Bone Marrow Function, Adequate Renal Function, Adequate Liver Function, Normal pancreatic function: amylase and lipase levels ≤ 1.5 x ULN. Blood pressure within upper limit of normal as defined below based on the average of the 2nd and 3rd of a total of 3 consecutive measurements, 5 minutes apart. Antihypertensives are permissible to achieve blood pressure within ULN, however must be on stable antihypertensive regimen with no adjustments within 14 days of enrollment.
8. Sexually active women of childbearing potential and fertile male participants and their partners must agree to use effective methods of contraception e.g., hormonal oral contraception, injectables, intrauterine device, surgical sterilization including vasectomy, or hormonal implant with barrier methods (male condom, female condom, or diaphragm with spermicidal gel) during the course of the study and for 4 months after the last dose of study treatment. Barrier methods alone are insufficient. True sexual abstinence or evidence of surgical sterility (e.g. vasectomized partner, post-hysterectomy, menopause with last menstrual period >=12 months prior to screening visit) are acceptable method of birth control. Persons of childbearing potential will be given a pregnancy test within 14 days prior to first dose of study treatment and must have a negative urine or serum pregnancy test.
9. The participant is not planning to undergo surgery or other interventions/ treatments for the target lesion, except protocol specified therapy, for the duration of the study.
10. The participant or the participant's legal authorized representative is able to understand the informed consent form describing the risks of the study and voluntarily signs the informed consent document.
11. In the opinion of the investigator, the participant is willing and able to attend study visits, comply with the study procedures as specified in the protocol, and comply with the administration of the study drug.

Exclusion Criteria:

1. Prior treatment with HLX-1502 for a PN.
2. The participant has used any of the following systemic medications/ therapies within the specified period prior to enrollment: MEK-inhibitors, other drugs in the TKI class, HLX-1502, Participants may have received treatment for a PN or other tumor/malignancy but must have fully recovered to baseline or CTCAE ≤ Grade 1 from acute toxicities from prior therapies except alopecia, Myelosuppressive chemotherapy, Hematopoietic growth factors, Biologic (anti-neoplastic agent), Investigational Drugs, Any other systemically administered anti-neoplastic agent and Radiation therapy.
3. Evidence of an NF1-related tumor such as optic pathway or other low-grade glioma, high-grade glioma, malignant peripheral nerve sheath tumor, or other cancer/tumor requiring treatment with chemotherapy, biologic therapy, surgery or radiation therapy.
4. Participants with high-grade glioma, malignant peripheral nerve sheath tumor, or other malignancy who received treatment in the last 12 months. Exceptions include basal cell carcinoma of the skin and squamous cell carcinoma of the skin that have undergone potentially curative therapy. If the investigator has any clinical concerns for ANNUBP/Atypical Neurofibroma or MPNST, a biopsy sample must be taken prior to study confirming eligibility.
5. Dental braces or prosthesis that interfere with volumetric analysis of the neurofibroma(s).
6. Surgery: Any major surgery within 12 weeks before starting the Treatment Period or foreseen during participation in the trial, any minor surgeries within 1 month before first dose of study treatment and Participants must have complete wound healing from major surgery or minor surgery before the first dose of study treatment. Participants with clinically relevant ongoing complications from prior surgery are not eligible.
7. Cataracts noted on ophthalmologic exam.
8. Cardiovascular disorders.
9. Other clinically significant disorders that would preclude safe study participation, including active infection, a known history of HIV seropositivity or known immunodeficiency or Known history of Hepatitis B or Hepatitis C.
10. Participants who require treatment with a drug that is a substrate of CYP1A2, CYP2C8, UGT1A1, UGT1A3 with a narrow therapeutic index during protocol therapy.
11. Known severe sensitivity to HLX-1502 or any excipient of HLX-1502 or history of allergic reactions attributed to compounds of similar chemical or biologic composition to HLX-1502.
12. Known severe sensitivity to FD&C Yellow No. 5.
13. Participants receiving therapeutic anticoagulation with vitamin K antagonist.
14. Participants presently with iron deficiency and/or actively receiving iron replacement or requiring treatment with copper or zinc for any indication at study baseline.
15. Pregnant or breast-feeding women.
16. Unable or unwilling to swallow tablets.
17. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter ingestion and/or the absorption of HLX-1502.
18. Participants who have other medical, social or concurrent challenges that are likely to negatively impact their ability to meet all of the trial obligations and therefore may increase the risk of safe participation in the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
PN response rate | 12 months
  Response will be determined by a blinded centralized review of volumetric MRI. A partial response (PR) is defined as ≥ 20% decrease in the volume of target PN.

SECONDARY OUTCOMES:
Duration of response (DOR) and Time to response (TOR) | 12 months
  Response will be determined by a blinded centralized review of volumetric MRI.
Safety and tolerability of HLX-1502 | 12 months
  Adverse events (AEs) will be assessed according to toxicities graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
PN response rate | 24 months
  Response will be determined by a blinded centralized review of volumetric MRI. A partial response (PR) is defined as ≥ 20% decrease in the volume of target PN.
Pharmacokinetics of HLX-1502 | 12 months
  Measured by plasma concentrations
Confirmed PN response rate | 12 and 24 months
  Confirmed response will be determined by a blinded centralized review of volumetric MRI

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Bornhorst, Study Chair — Lurie's Children's Hospital; Michael Fisher, Study Chair — Children's Hospital of Philadelphia; Kathryn Nevel, Study Chair — Indiana University
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - New York University Langone Health, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No